CLINICAL TRIAL: NCT00304577
Title: A Randomized Comparison of Bilateral Recession With Unilateral Recession-Resection as Surgery for Infantile Esotropia
Brief Title: Bilateral Recession or Unilateral Recession-Resection as Surgery for Infantile Esotropia
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Other Study IDs: 662720
Record Dates: First submitted 2006-03-17; First posted 2006-03-20 (Estimated); Last update posted 2006-03-20 (Estimated); Status verified 2005-09

CONDITIONS: Strabismus
Keywords: Strabismus; Esotropia; Surgical techniques
MeSH Terms: conditions — Strabismus; Esotropia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Bilateral recession
Procedure: Unilateral recession and resection

SUMMARY:
Infantile esotropia is corrected in most cases by bilateral recession of the medial rectus muscles (BR) or by unilateral recession of the medial rectus muscle and resection of the lateral rectus muscle (RR). We compared the outcome of these techniques in a randomized prospective study.

DETAILED DESCRIPTION:
We randomly assigned 124 patients (average age 5.8) from twelve participating clinics in Germany and the Netherlands to either BR or RR. Patients did not have demonstrable binocular vision at baseline. The angle of strabismus was measured pre- and postoperatively in a standardized fashion. The primary parameter to assess difference between BR and RR was the variation of the latent angle of strabismus at distance at three months postoperatively, secondary outcomes were reduction of convergence excess and binocular vision.

ELIGIBILITY:
Inclusion Criteria:

* Eligible were all children aged three to eight years with a normal psychophysical development, and onset of esotropia before age one who visited one of the clinics during the study period.

Exclusion Criteria:

* previous strabismus surgery, an angle of strabismus larger than 24° or smaller than 10°, any normal binocular vision, convergence excess with angle of strabismus at near fixation 1.5 times larger than the angle at distance, more than 1 line Logmar acuity difference between the two eyes, hypermetropia over 6 diopters or myopia over 3 diopters, up- or downshoot in (25°) adduction more than 8°, V-pattern (25° up and down gaze) over 8°, A-pattern (25° up and down gaze) over 5° and manifest vertical strabismus over 4°

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Dates: Start 1998-01; Study Completion 2001-12

CONTACTS AND LOCATIONS:
Overall Officials: Huib J. Simonsz, MD, PhD, Study Chair — Erasmus MC, Rotterdam
Locations (12):
- Germany (9):
  - Dept. Ophthalmology, Bonn
  - Dept. Ophthalmology, Erlangen
  - Dept. Ophthalmology, Essen
  - Dept. Ophthalmology, Frankfurt
  - Dept. Ophthalmology, Freiburg im Breisgau
  - Dept. Ophthalmology, Hamburg
  - Dept. Ophthalmology, Heidelberg
  - Dept. Ophthalmology, Regensburg
  - Dept. Ophthalmology, Tübingen
- Netherlands (3):
  - Dept. Ophthalmology, Maastricht
  - Erasmus MC, Rotterdam
  - Dept. Ophthalmology, Utrecht